CLINICAL TRIAL: NCT06601842
Title: Monitoring and Optimization of Cerebral Perfusion Pressure in Post-cardiac Arrest Patients: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202407092RINE
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; post-arrest care; ICP monitor; Cerebral perfusion pressure
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP monitoring (Experimental): ICP monitoring
  Interventions: Device: ICP monitoring

INTERVENTIONS:
Device: ICP monitoring — ICP monitoring

SUMMARY:
The goal of this study is to establish the ICP and CPP monitoring process and analyze the results in post-arrest patients, to validate the correlation between direct and non-invasive ICP monitoring indicators, to establish a protocol of management of elevated ICP and insufficient CPP in post-arrest care, to establish a protocol for personalizing CPP and MAP optimization, and to analyze its impact on neuroprognosis.

Participants will receive ICP monitoring within 12 hours post-ROSC if meet all inclusion and exclusion criteria.

DETAILED DESCRIPTION:
Post-resuscitation care after cardiac arrest is an important emergency and critical care issue. The post-arrest care after the return of spontaneous circulation has also been incorporated into the chain of survival and resuscitation guidelines. After the regain of spontaneous circulation, cardiac arrest patients will face the challenges of post-arrest syndrome, which includes post-anoxic brain injury, myocardial dysfunction, systemic ischemia-reperfusion, and persistent precipitating causes. The hypoxic brain injury will impair the autoregulation of cerebral blood vessels, thereby affecting the adjustment of intracranial pressure (ICP) and causing cerebral edema. High-quality post-arrest care including targeted temperature management, optimization of hemodynamics and respiratory care, control of blood sugar, monitoring and treatment of epilepsy, etc. The goal is to achieve neuroprotective effects and improve patient outcomes.

The modalities that currently have more evidence for neurocritical care and neuroprognosis include electroencephalogram (EEG) monitoring, pupillary light reflex, brain imaging such as computed tomography (CT) and magnetic resonance imaging (MRI), somatosensory evoked potentials (SSEP), and serum biomarkers such as neuron-specific enolase (NSE), etc. Direct ICP monitoring is not routinely used in cardiac arrest patients due to a lack of clinical experience and concurrent use of antiplatelet medications or anticoagulants. The application of ICP monitoring in neurocritical care can be based on the experience of traumatic brain injury. ICP monitoring can facilitate early detection, determination of treatment strategies, and prediction of outcomes. Cerebral perfusion pressure (CPP) can also be obtained by ICP monitoring. Current head injury treatment guidelines recommend maintaining CPP at around 60-70 mmHg. However, there are no current recommendations for CPP standards for post-arrest patients. In recent years, there have been studies on the utilization of the pressure reactivity index to identify the optimized CPP in patients with traumatic brain injury, but not yet applicated in post-arrest patients.

This study aims to establish the ICP and CPP monitoring process and analyze the result in post-arrest patients, to validate the correlation between direct and non-invasive ICP monitoring indicators, to establish a protocol of management of elevated ICP and insufficient CPP in post-arrest care, to establish a protocol for personalizing CPP and MAP optimization, and to analyze its impact on neuroprognosis.

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic cardiac arrest
* admitted to ICU
* GCS: motor <=5
* severity: TIMECARD score medium-risk group

Exclusion Criteria:

* traumatic cardiac arrest
* pregnancy
* intracranial hemorrhage
* coagulopathy
* anti-platelet or anti-coagulation use
* terminal illness
* pre-arrest CPC score >=3
* GWR < 1.2 on CT or severe hypoxic ischemic encephalopathy
* CNS infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ICP difference between different temperature | 12 hour, day 1, 3, 7 post-ROSC

SECONDARY OUTCOMES:
Difference between direct and non-invasive ICP monitoring indicators | 12 hour, day 1, 3, 7 post-ROSC

CONTACTS AND LOCATIONS:
Overall Officials: Dean-An Ling, MD, Study Director — National Taiwan University Medical College and Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyckoff MH, Greif R, Morley PT, Ng KC, Olasveengen TM, Singletary EM, Soar J, Cheng A, Drennan IR, Liley HG, Scholefield BR, Smyth MA, Welsford M, Zideman DA, Acworth J, Aickin R, Andersen LW, Atkins D, Berry DC, Bhanji F, Bierens J, Borra V, Bottiger BW, Bradley RN, Bray JE, Breckwoldt J, Callaway CW, Carlson JN, Cassan P, Castren M, Chang WT, Charlton NP, Chung SP, Considine J, Costa-Nobre DT, Couper K, Couto TB, Dainty KN, Davis PG, de Almeida MF, de Caen AR, Deakin CD, Djarv T, Donnino MW, Douma MJ, Duff JP, Dunne CL, Eastwood K, El-Naggar W, Fabres JG, Fawke J, Finn J, Foglia EE, Folke F, Gilfoyle E, Goolsby CA, Granfeldt A, Guerguerian AM, Guinsburg R, Hirsch KG, Holmberg MJ, Hosono S, Hsieh MJ, Hsu CH, Ikeyama T, Isayama T, Johnson NJ, Kapadia VS, Kawakami MD, Kim HS, Kleinman M, Kloeck DA, Kudenchuk PJ, Lagina AT, Lauridsen KG, Lavonas EJ, Lee HC, Lin YJ, Lockey AS, Maconochie IK, Madar RJ, Malta Hansen C, Masterson S, Matsuyama T, McKinlay CJD, Meyran D, Morgan P, Morrison LJ, Nadkarni V, Nakwa FL, Nation KJ, Nehme Z, Nemeth M, Neumar RW, Nicholson T, Nikolaou N, Nishiyama C, Norii T, Nuthall GA, O'Neill BJ, Ong YG, Orkin AM, Paiva EF, Parr MJ, Patocka C, Pellegrino JL, Perkins GD, Perlman JM, Rabi Y, Reis AG, Reynolds JC, Ristagno G, Rodriguez-Nunez A, Roehr CC, Rudiger M, Sakamoto T, Sandroni C, Sawyer TL, Schexnayder SM, Schmolzer GM, Schnaubelt S, Semeraro F, Skrifvars MB, Smith CM, Sugiura T, Tijssen JA, Trevisanuto D, Van de Voorde P, Wang TL, Weiner GM, Wyllie JP, Yang CW, Yeung J, Nolan JP, Berg KM; Collaborators. 2022 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations: Summary From the Basic Life Support; Advanced Life Support; Pediatric Life Support; Neonatal Life Support; Education, Implementation, and Teams; and First Aid Task Forces. Circulation. 2022 Dec 20;146(25):e483-e557. doi: 10.1161/CIR.0000000000001095. Epub 2022 Nov 3. PMID 36325905
- [Background] Kirkegaard H, Taccone FS, Skrifvars M, Soreide E. Postresuscitation Care after Out-of-hospital Cardiac Arrest: Clinical Update and Focus on Targeted Temperature Management. Anesthesiology. 2019 Jul;131(1):186-208. doi: 10.1097/ALN.0000000000002700. PMID 31021845
- [Background] Nolan JP, Soar J, Cariou A, Cronberg T, Moulaert VR, Deakin CD, Bottiger BW, Friberg H, Sunde K, Sandroni C. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines for Post-resuscitation Care 2015: Section 5 of the European Resuscitation Council Guidelines for Resuscitation 2015. Resuscitation. 2015 Oct;95:202-22. doi: 10.1016/j.resuscitation.2015.07.018. No abstract available. PMID 26477702
- [Background] Neumar RW, Nolan JP, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT Jr, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation (American Heart Association, Australian and New Zealand Council on Resuscitation, European Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Asia, and the Resuscitation Council of Southern Africa); the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; and the Stroke Council. Circulation. 2008 Dec 2;118(23):2452-83. doi: 10.1161/CIRCULATIONAHA.108.190652. Epub 2008 Oct 23. No abstract available. PMID 18948368
- [Background] Nolan JP, Sandroni C, Bottiger BW, Cariou A, Cronberg T, Friberg H, Genbrugge C, Haywood K, Lilja G, Moulaert VRM, Nikolaou N, Olasveengen TM, Skrifvars MB, Taccone F, Soar J. European Resuscitation Council and European Society of Intensive Care Medicine guidelines 2021: post-resuscitation care. Intensive Care Med. 2021 Apr;47(4):369-421. doi: 10.1007/s00134-021-06368-4. Epub 2021 Mar 25. PMID 33765189
- [Background] Sandroni C, Skrifvars MB, Taccone FS. Brain monitoring after cardiac arrest. Curr Opin Crit Care. 2023 Apr 1;29(2):68-74. doi: 10.1097/MCC.0000000000001023. Epub 2023 Feb 16. PMID 36762679
- [Background] Gueugniaud PY, Garcia-Darennes F, Gaussorgues P, Bancalari G, Petit P, Robert D. Prognostic significance of early intracranial and cerebral perfusion pressures in post-cardiac arrest anoxic coma. Intensive Care Med. 1991;17(7):392-8. doi: 10.1007/BF01720676. PMID 1774392
- [Background] Sekhon MS, Griesdale DE, Ainslie PN, Gooderham P, Foster D, Czosnyka M, Robba C, Cardim D. Intracranial pressure and compliance in hypoxic ischemic brain injury patients after cardiac arrest. Resuscitation. 2019 Aug;141:96-103. doi: 10.1016/j.resuscitation.2019.05.036. Epub 2019 Jun 8. PMID 31185256
- [Background] Kjaergaard J, Moller JE, Schmidt H, Grand J, Molstrom S, Borregaard B, Veno S, Sarkisian L, Mamaev D, Jensen LO, Nyholm B, Hofsten DE, Josiassen J, Thomsen JH, Thune JJ, Obling LER, Lindholm MG, Frydland M, Meyer MAS, Winther-Jensen M, Beske RP, Frikke-Schmidt R, Wiberg S, Boesgaard S, Madsen SA, Jorgensen VL, Hassager C. Blood-Pressure Targets in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Oct 20;387(16):1456-1466. doi: 10.1056/NEJMoa2208687. Epub 2022 Aug 27. PMID 36027564
- [Background] Tas J, Beqiri E, van Kaam RC, Czosnyka M, Donnelly J, Haeren RH, van der Horst ICC, Hutchinson PJ, van Kuijk SMJ, Liberti AL, Menon DK, Hoedemaekers CWE, Depreitere B, Smielewski P, Meyfroidt G, Ercole A, Aries MJH. Targeting Autoregulation-Guided Cerebral Perfusion Pressure after Traumatic Brain Injury (COGiTATE): A Feasibility Randomized Controlled Clinical Trial. J Neurotrauma. 2021 Oct 15;38(20):2790-2800. doi: 10.1089/neu.2021.0197. Epub 2021 Aug 16. PMID 34407385
- [Background] Tsigaras ZA, Weeden M, McNamara R, Jeffcote T, Udy AA; PRECISION-TBI Investigators. The pressure reactivity index as a measure of cerebral autoregulation and its application in traumatic brain injury management. Crit Care Resusc. 2023 Dec 14;25(4):229-236. doi: 10.1016/j.ccrj.2023.10.009. eCollection 2023 Dec. PMID 38234328